CLINICAL TRIAL: NCT02387996
Title: A Phase II Single Arm Clinical Trial of Nivolumab (BMS-936558) in Subjects With Metastatic or Unresectable Urothelial Cancer Who Have Progressed or Recurred Following Treatment With a Platinum Agent
Brief Title: A Study of Nivolumab in Participants With Metastatic or Unresectable Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-275
Record Dates: First submitted 2015-02-26; First posted 2015-03-13 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Various Advanced Cancer
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab intravenous infusion as specified
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab
  Other Names: BMS(936558)

SUMMARY:
The purpose the study is to measure the effect of nivolumab (BMS-936558) in reducing tumor size in subjects with metastatic or unresectable bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of metastatic or surgically unresectable transitional cell carcinoma of the urothelium involving the bladder,urethra,ureter or renal pelvis
* Measurable disease by CT or MRI
* Progression or recurrence after treatment
* i) With at least 1 platinum-containing chemotherapy regimen for metastatic or surgically unresectable locally advanced urothelial cancer, or
* ii) Within 12 months of peri-operative (neo-adjuvant or adjuvant) treatment with a platinum agent in the setting of cystectomy for localized muscle-invasive urothelial cancer
* Subject that have received more than 2 prior lines of chemotherapy must not have liver metastases
* Tumor tissues (archived or new biopsy) must be provided for biomarker analysis
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1

Exclusion Criteria:

* Subjects with active cancer that has spread to the central nervous system
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured
* Subject with active, known or suspected autoimmune disease
* Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 day of study drug administration
* Prior treatment with an anti-PD-1,anti-PD-L1,anti-PD-L2,anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody, anti-CD137 or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways

Exclusion laboratory criteria:

* Positive test for hepatitis B virus surface antigen (HBV s Ag) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Known history of testing positive for human Immunodeficiency virus (HIV) or known acquired Immunodeficiency syndrome (AIDS)

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2021-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (67):
- United States (19):
  - Local Institution - 0013, Phoenix, Arizona
  - Local Institution - 0012, Duarte, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Local Institution - 0016, Aurora, Colorado
  - University Cancer Blood Ctr, Athens, Georgia
  - Ft. Wayne Med Onco-Hema Inc, Fort Wayne, Indiana
  - Local Institution - 0030, Indianapolis, Indiana
  - Local Institution - 0052, Iowa City, Iowa
  - Crescent City Research Consortium, LLC, Marrero, Louisiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - GU Research Network, LLC, Omaha, Nebraska
  - Local Institution - 0028, New York, New York
  - Local Institution - 0004, Charlotte, North Carolina
  - Local Institution - 0051, Portland, Oregon
  - Local Institution - 0029, Philadelphia, Pennsylvania
  - Local Institution - 0059, Pittsburgh, Pennsylvania
  - Erlanger Oncology & Hematology - Univ. of TN, Chattanooga, Tennessee
  - Local Institution - 0001, Houston, Texas
  - Local Institution - 0036, Seattle, Washington
- Australia (2):
  - Local Institution - 0060, Waratah, New South Wales
  - Local Institution - 0070, Elizabeth Vale, South Australia
- Belgium (3):
  - Local Institution - 0022, Brussels
  - Local Institution - 0023, Edegem
  - Local Institution - 0024, Hasselt
- Czechia (3):
  - Local Institution - 0027, Brno
  - Local Institution - 0026, Olomouc
  - Local Institution, Prague
- Finland (2):
  - Local Institution - 0010, Helsinki
  - Local Institution - 0009, Tampere
- Germany (8):
  - Local Institution - 0049, Erfurt
  - Local Institution - 0047, Erlangen
  - Local Institution - 0042, Hamburg
  - Local Institution - 0043, Heidelberg
  - Local Institution - 0015, Jena
  - Local Institution - 0041, München
  - Local Institution, Rostock
  - Local Institution - 0048, Tübingen
- Italy (5):
  - Local Institution - 0017, Arezzo
  - Local Institution - 0020, Milan
  - Local Institution - 0018, Napoli
  - Local Institution - 0050, Pavia
  - Local Institution - 0021, Roma
- Japan (14):
  - Local Institution - 0074, Akita, Akita
  - Local Institution - 0083, Hirosaki-shi, Aomori
  - Local Institution - 0081, Tsukuba, Ibaraki
  - Local Institution - 0078, Morioka, Iwate
  - Local Institution, Yokohama, Kanagawa
  - Local Institution - 0080, Kumamoto, Kumamoto
  - Local Institution - 0082, Kyoto, Kyoto
  - Local Institution - 0076, Niigata, Niigata
  - Local Institution - 0084, Osaka-Sayama-Shi, Osaka
  - Local Institution - 0085, Bunkyo-ku, Tokyo
  - Local Institution - 0073, Bunkyo-ku, Tokyo
  - Local Institution - 0077, Bunkyo-ku, Tokyo
  - Local Institution - 0086, Shinjuku-ku, Tokyo
  - Local Institution - 0075, Shinjuku-ku, Tokyo
- Poland (5):
  - Local Institution, Gdansk
  - Local Institution - 0046, Krakow
  - Local Institution - 0040, Lodz
  - Local Institution - 0056, Szczecin
  - Local Institution - 0038, Wroclaw
- Spain (5):
  - Local Institution - 0035, Badalona-barcelona
  - Local Institution - 0033, Barcelona
  - Local Institution - 0034, Hospitalet de Llobregat - Barcelona
  - Local Institution - 0031, Madrid
  - Local Institution - 0032, Seville
- Local Institution - 0014, Lund, Sweden

REFERENCES:
- [Derived] Sharma P, Retz M, Siefker-Radtke A, Baron A, Necchi A, Bedke J, Plimack ER, Vaena D, Grimm MO, Bracarda S, Arranz JA, Pal S, Ohyama C, Saci A, Qu X, Lambert A, Krishnan S, Azrilevich A, Galsky MD. Nivolumab in metastatic urothelial carcinoma after platinum therapy (CheckMate 275): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2017 Mar;18(3):312-322. doi: 10.1016/S1470-2045(17)30065-7. Epub 2017 Jan 26. PMID 28131785
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab 3 mg/kg: Nivolumab 3 mg/kg was administered as a 60 minute IV infusion Q2W
Period: Overall Study
Arm/Group | Nivolumab 3 mg/kg
Started | 270
Completed (Completed=continuing in the study treatment) | 0
Not Completed | 270
Not completed — Disease Progression | 167
Not completed — Study Drug Toxicity | 31
Not completed — Adverse Event Unrelated to Study Drug | 39
Not completed — Participant Request to Discontinue Treatment | 20
Not completed — Subject Withdrew Consent | 5
Not completed — Lost to Follow-up | 1
Not completed — Poor/Non-Compliance | 1
Not completed — Other Reasons | 5
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: All Treated Participants
Arm/Group | Nivolumab 3 mg/kg
Number analyzed (Participants) | 270
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 211
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 156
  Unknown or Not Reported | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 231
  Black or African American | 2
  Asian | 30
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Other | 3
  Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Per BIRC Assessment
Description: Objective Response Rate (ORR) was defined as the number of participants with a best overall response of confirmed Complete Response (CR) or Partial Response (PR) (per RECIST 1.1 criteria) divided by the number of all treated participants. RECIST 1.1 = Response Evaluation Criteria in Solid Tumors. CR= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. BIRC= blinded independent review committee
Time Frame: From the date of first dose to the date of objectively documented progression or the date of subsequent therapy, whichever occurs first (assessed up to 14 months)
Population: All treated participants. Treated participants from Japan enrolled after main enrollment period were excluded from primary efficacy analysis.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Nivolumab 3 mg/kg
Number analyzed (Participants) | 265
Percent of participants | 19.6 [15.0 to 24.9]

2. Primary Outcome: ORR Per BIRC Assessment by PD-L1 Expression Level
Description: Objective Response Rate (ORR) was defined as the number of participants with a best overall response of confirmed Complete Response (CR) or Partial Response (PR) (per RECIST 1.1 criteria) divided by the number of all treated participants. RECIST 1.1 = Response Evaluation Criteria in Solid Tumors. CR= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. BIRC= blinded independent review committee PD-L1 expression level= membranous staining in greater than or equal to 5% and greater than or equal to 1% tumor cells. n = Number of participants in each category
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Nivolumab 3 mg/kg
Number analyzed (Participants) | 265
Percent of Participants
  PD-L1 <1% | 16.1 [10.5 to 23.1]
  PD-L1 >= 1% | 23.8 [16.5 to 32.3]
  PD-L1 <5% | 15.8 [10.8 to 21.8]
  PD-L1 >=5% | 28.4 [18.9 to 39.5]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from first dosing date to the date of the first documented tumor progression, based on Blinded Independent Review Committee (BIRC) assessments or death due to any cause. Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. PD-L1 expression level is defined as membranous staining in greater than or equal to 5% and greater than or equal to 1% tumor cells.
Time Frame: From first dosing date to the date of the first documented tumor progression (up to approximately 6 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3 mg/kg
Number analyzed (Participants) | 270
Months
  All treated participants | 1.94 [1.87 to 2.33]
  PD-L1 <1%: number analyzed (Participants) | 146
  PD-L1 <1% | 1.87 [1.74 to 2.00]
  PD-L1 >= 1%: number analyzed (Participants) | 124
  PD-L1 >= 1% | 3.45 [1.91 to 3.71]
  PD-L1 <5%: number analyzed (Participants) | 187
  PD-L1 <5% | 1.87 [1.81 to 2.04]
  PD-L1 >=5%: number analyzed (Participants) | 83
  PD-L1 >=5% | 3.68 [1.91 to 5.52]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time from first dosing date to the date of death. A participant who had not died was censored at last known date alive. PD-L1 expression level = membranous staining in greater than or equal to 5% and greater than or equal to 1% tumor cells.
Time Frame: From first dosing date to the date of death (up to approximately 23 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3 mg/kg
Number analyzed (Participants) | 270
Months
  All treated participants | 8.57 [6.05 to 11.27]
  PD-L1 <1%: number analyzed (Participants) | 146
  PD-L1 <1% | 5.95 [4.37 to 8.08]
  PD-L1 >= 1%: number analyzed (Participants) | 124
  PD-L1 >= 1% | 11.86 [9.10 to 19.12]
  PD-L1 <5%: number analyzed (Participants) | 187
  PD-L1 <5% | 6.24 [4.96 to 9.00]
  PD-L1 >=5%: number analyzed (Participants) | 83
  PD-L1 >=5% | 13.54 [9.63 to 22.14]

5. Secondary Outcome: Objective Response Rate (ORR) Per Investigator
Description: Investigator-assessed ORR was defined as the percent of participants with a best overall response of confirmed complete response (CR) or partial response (PR). Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD-L1 expression level = Membranous staining in greater than or equal to 5% and greater than or equal to 1% tumor cells.
Time Frame: From the date of first dose to the date of objectively documented progression or the date of subsequent therapy, whichever occurs first (up to approximately 45 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Nivolumab 3 mg/kg
Number analyzed (Participants) | 270
Percent of Participants
  All treated participants | 24.8 [19.8 to 30.4]
  PD-L1 <1%: number analyzed (Participants) | 146
  PD-L1 <1% | 19.9 [13.7 to 27.3]
  PD-L1 >= 1%: number analyzed (Participants) | 124
  PD-L1 >= 1% | 30.6 [22.7 to 39.6]
  PD-L1 <5%: number analyzed (Participants) | 187
  PD-L1 <5% | 20.9 [15.3 to 27.4]
  PD-L1 >=5%: number analyzed (Participants) | 83
  PD-L1 >=5% | 33.7 [23.7 to 44.9]

6. Post Hoc Outcome: Time to Response (TTR) - Extended Collection
Description: TTR is defined as the time from first dosing date to the date of the first confirmed complete response (CR) or partial response (PR), as assessed by the Blinded Independent Review Committee (BIRC). Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Note: This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date.
Time Frame: From first dosing date to the date of the first confirmed response (up to approximately 14 months)
Population: All responders-includes responders who had neither progressed nor initiated subsequent therapy at the time of analysis, and excludes responders censored prior to 12 weeks of the clinical data cutoff date (if this cutoff date is before week 48) or prior to 18 weeks of the clinical data cutoff date (if this cutoff date is after or on week 48)
Measure: Median (Full Range); unit: Months
Arm/Group | Nivolumab 3 mg/kg
Number analyzed (Participants) | 56
Months | 1.97 [1.6 to 13.8]

7. Post Hoc Outcome: Duration of Response (DOR) - Extended Collection
Description: DOR is the time from first confirmed response, complete (CR) or partial response (PR) to the date of the first tumor progression PER RECIST 1.1 criteria or death due to any cause, whichever occurs first. Participants without prior reported progression will be censored at the last evaluable tumor assessments prior to subsequent anticancer therapy. Participants who die without a reported prior progression will be considered on the date of their death. Participants who neither progress nor die will be censored on the date of their last evaluable tumor assessment. CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions. Note: This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date.
Time Frame: From the first confirmed response to the date of the first documented tumor progression or death due to any cause, whichever occurs first (up to approximately 32 months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3 mg/kg
Number analyzed (Participants) | 56
Months | 20.27 [11.50 to 31.31]

8. Primary Outcome: Time to Response (TTR)
Description: TTR is defined as the time from first dosing date to the date of the first confirmed complete response (CR) or partial response (PR), as assessed by the Blinded Independent Review Committee (BIRC). Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dosing date to the date of the first confirmed response (up to approximately 14 months)
Population: as for outcome 6
Measure: Median (Full Range); unit: Months
Arm/Group | Nivolumab 3 mg/kg
Number analyzed (Participants) | 52
Months | 1.87 [1.6 to 5.9]

9. Primary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from first confirmed response, complete response (CR) or partial response (PR) to the date of the first documented tumor progression as determined using RECIST 1.1 criteria or death due to any cause, whichever occurs first. Participants who start subsequent therapy without a prior reported progression will be censored at the last evaluable tumor assessments prior to initiation of the subsequent anticancer therapy. Participants who die without a reported prior progression will be considered to have progressed on the date of their death. Participants who neither progress nor die will be censored on the date of their last evaluable tumor assessment.
Time Frame: From the first confirmed response to the date of the first documented tumor progression or death due to any cause, whichever occurs first (up to approximately 14 months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3 mg/kg
Number analyzed (Participants) | 52
Months | NA [7.43 to NA] — Median and upper limit not calculated due to insufficient number of events.

10. Post Hoc Outcome: Objective Response Rate (ORR) Per BIRC Assessment - Extended Collection
Description: Objective Response Rate (ORR) was defined as the percent of participants with a best overall response of confirmed Complete Response (CR) or Partial Response (PR) (per RECIST 1.1 criteria). RECIST 1.1 = Response Evaluation Criteria in Solid Tumors. CR= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. BIRC= blinded independent review committee PD-L1 expression level= membranous staining in greater than or equal to 5% and greater than or equal to 1% tumor cells.
  Note: This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date."
Time Frame: From the date of first dose to the date of objectively documented progression or the date of subsequent therapy, whichever occurs first (up approximately to 43 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Nivolumab 3 mg/kg
Number analyzed (Participants) | 270
Percent of Participants
  All treated participants | 20.7 [16.1 to 26.1]
  PD-L1 <1%: number analyzed (Participants) | 146
  PD-L1 <1% | 16.4 [10.8 to 23.5]
  PD-L1 >= 1%: number analyzed (Participants) | 124
  PD-L1 >= 1% | 25.8 [18.4 to 34.4]
  PD-L1 <5%: number analyzed (Participants) | 187
  PD-L1 <5% | 16.0 [11.1 to 22.1]
  PD-L1 >=5%: number analyzed (Participants) | 83
  PD-L1 >=5% | 31.3 [21.6 to 42.4]

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to study completion, (up to approximately 80 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 78 months).
Arm/Group | Nivolumab 3 mg/kg
All-Cause Mortality (participants affected / at risk) | 225/270
Serious Adverse Events (participants affected / at risk) | 199/270
Other Adverse Events (participants affected / at risk) | 245/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg (N=270)
Agranulocytosis (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Atrial flutter (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Hypertensive heart disease (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 3
Hypophysitis (Endocrine disorders) | 1
Uveitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 1
Autoimmune colitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 7
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2
Duodenitis (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 4
Intestinal perforation (Gastrointestinal disorders) | 3
Large intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 2
Disease progression (General disorders) | 1
Fatigue (General disorders) | 3
General physical health deterioration (General disorders) | 12
Malaise (General disorders) | 2
Mass (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Obstruction (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 5
Pelvic mass (General disorders) | 1
Pyrexia (General disorders) | 4
Sudden death (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Biliary obstruction (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 3
Anal abscess (Infections and infestations) | 1
Arthritis infective (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Candida infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Clostridium difficile infection (Infections and infestations) | 1
Coronavirus infection (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Infected lymphocele (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 12
Septic shock (Infections and infestations) | 4
Staphylococcal infection (Infections and infestations) | 1
Stoma site cellulitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 17
Urosepsis (Infections and infestations) | 3
Femur fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Blood bilirubin increased (Investigations) | 3
Hepatic enzyme increased (Investigations) | 1
Influenza A virus test positive (Investigations) | 1
Lipase increased (Investigations) | 1
Liver function test increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Quality of life decreased (Investigations) | 1
Transaminases increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 95
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell cancer of renal pelvis and ureter metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Brain oedema (Nervous system disorders) | 2
Cerebellar haematoma (Nervous system disorders) | 1
Cerebral disorder (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Epilepsy (Nervous system disorders) | 2
Monoplegia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Device dislocation (Product Issues) | 1
Thrombosis in device (Product Issues) | 1
Anxiety (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Bladder tamponade (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 4
Hydronephrosis (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Pemphigoid (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Arteriovenous fistula (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 4
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg (N=270)
Anaemia (Blood and lymphatic system disorders) | 58
Hypothyroidism (Endocrine disorders) | 32
Abdominal pain (Gastrointestinal disorders) | 34
Constipation (Gastrointestinal disorders) | 60
Diarrhoea (Gastrointestinal disorders) | 60
Nausea (Gastrointestinal disorders) | 71
Vomiting (Gastrointestinal disorders) | 42
Asthenia (General disorders) | 43
Chills (General disorders) | 22
Fatigue (General disorders) | 97
Oedema peripheral (General disorders) | 45
Pyrexia (General disorders) | 65
Nasopharyngitis (Infections and infestations) | 16
Upper respiratory tract infection (Infections and infestations) | 20
Urinary tract infection (Infections and infestations) | 43
Amylase increased (Investigations) | 20
Blood alkaline phosphatase increased (Investigations) | 14
Blood creatinine increased (Investigations) | 24
Lipase increased (Investigations) | 18
Weight decreased (Investigations) | 24
Decreased appetite (Metabolism and nutrition disorders) | 74
Dehydration (Metabolism and nutrition disorders) | 21
Hyperglycaemia (Metabolism and nutrition disorders) | 16
Hypokalaemia (Metabolism and nutrition disorders) | 15
Hyponatraemia (Metabolism and nutrition disorders) | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 40
Back pain (Musculoskeletal and connective tissue disorders) | 41
Bone pain (Musculoskeletal and connective tissue disorders) | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25
Dizziness (Nervous system disorders) | 21
Headache (Nervous system disorders) | 20
Paraesthesia (Nervous system disorders) | 14
Anxiety (Psychiatric disorders) | 17
Insomnia (Psychiatric disorders) | 29
Haematuria (Renal and urinary disorders) | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 59
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 45
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 15
Dry skin (Skin and subcutaneous tissue disorders) | 16
Pruritus (Skin and subcutaneous tissue disorders) | 45
Rash (Skin and subcutaneous tissue disorders) | 46
Hypotension (Vascular disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.